CLINICAL TRIAL: NCT03270332
Title: Effect of Inhaled Albuterol on Pulmonary Hemodynamics in Patients With Group 1 Pulmonary Arterial Hypertension on Oral Pulmonary Vasodilator Therapy: A Proof of Concept Study
Brief Title: Effect of Inhaled Albuterol in Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20170552
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albuterol followed by placebo (Experimental): Participants in this group will receive albuterol first followed by Placebo on the next visit
  Interventions: Drug: Albuterol; Drug: Placebo
- Placebo followed by albuterol (Experimental): Participants in this group will receive placebo first followed by albuterol on the next visit
  Interventions: Drug: Albuterol; Drug: Placebo

INTERVENTIONS:
Drug: Albuterol — inhalation of 270μg albuterol through a spacer
Drug: Placebo — inhalation of placebo through a spacer

SUMMARY:
The purpose of the present pilot study is to test the hypothesis that in patients with group 1 pulmonary arterial hypertension (PAH) who are on regular oral pulmonary vasodilator therapy, inhaled albuterol causes transient pulmonary vasodilation.

ELIGIBILITY:
Inclusion Criteria:

* A Mean Pulmonary Artery Pressure >25mmHg, Pulmonary Vascular Resistance >3 wood/units and pulmonary arterial wedge pressure <15mmHg, as documented by right heart catheterization within the last 3 years
* Regular use of oral pulmonary vasodilators

Exclusion Criteria:

* Presence of chronic respiratory disease (as documented by prior lung imaging and pulmonary function tests), cardiovascular disease (as documented by prior echocardiography and/or left heart catheterization), thromboembolic PAH (as documented by pulmonary angiography)
* women of childbearing potential who do not use accepted birth- control measures
* pregnant and breast-feeding women
* respiratory infection within 4 weeks of testing
* A systemic systolic arterial BP> 150 and/or diastolic arterial BP>100 on the experiment day
* A resting O2 saturation of < 90%
* Current smoking
* BMI >35 kg/m2 and/or a diagnosis of obstructive sleep apnea
* Use of inhaled or intravenous pulmonary vasodilators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Albuterol Followed by Placebo | Placebo Followed by Albuterol
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol Followed by Placebo | Placebo Followed by Albuterol | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Pulmonary Artery Pressure (MPAP)
Description: Change in MPAP will be measured using echocardiogram
Time Frame: Baseline, up to 30 minutes after inhalation
Population: This is a cross-over study design. All enrolled participants received both the albuterol and placebo intervention.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Albuterol Group: This is a cross-over study design. All participants received albuterol
- Placebo Group: This is a cross-over design. All participants received placebo.
Arm/Group | Albuterol Group | Placebo Group
Number analyzed (Participants) | 9 | 9
mmHg | 6.5 (2.8) | 4.3 (3.0)

2. Secondary Outcome: Change in Pulmonary Vascular Resistance (PVR)
Description: Change in PVR will be measured using echocardiogram
Time Frame: Baseline, up to 30 minutes after inhalation
Population: This is a cross-over study design. All enrolled participants received both the albuterol and placebo intervention.
Measure: Mean (Standard Error); unit: dyn.s.cm-5
Groups:
- Albuterol Group: This is a cross-over study. All participants received albuterol.
- Placebo Group: This is a cross-over study. All participants received placebo.
Arm/Group | Albuterol Group | Placebo Group
Number analyzed (Participants) | 9 | 9
dyn.s.cm-5 | 217 (92) | 108 (153)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Albuterol Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03270332/Prot_SAP_000.pdf